CLINICAL TRIAL: NCT03220243
Title: A Phase I Study of Autologous Mesenchymal Stromal Cell Coated Fistula Plug in Patients With Rectovaginal Fistulizing Crohn's Disease
Brief Title: Stem Cell Coated Fistula Plug in Patients With Crohn's RVF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Eric J. Dozois, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-002892
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Fistula Vagina; Crohn Disease
MeSH Terms: conditions — Vaginal Fistula; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MSC-AFP Single Treatment Group (Experimental): Eligible patients will be treated, single treatment group, no placebo arm.
  Interventions: Drug: MSC-AFP

INTERVENTIONS:
Drug: MSC-AFP — Eligible patients will be treated with a fistula plug that has been coated with autologous mesenchymal stromal cells.
  Other Names: • mesenchymal stromal cell coated fistula plug

SUMMARY:
The purpose of this study is to determine the safety of using an autologous mesenchymal stromal cell (MSC) coated fistula plug in people with rectovaginal fistulizing Crohn's disease. This is an autologous product derived from the patient and used only for the same patient. Participants will be in this study for two years. There is potential to continue to monitor participants' progress with regular visits as part of standard of care. All study visits take place at Mayo Clinic and Rochester, MN.

The study visit schedule is as follows:

Visit 1 (Week -6) - Screening visit: exam under anesthesia and surgery to assess eligibility of fistula tract, take fat biopsy, if eligible, and fecal diversion.

Visit 2 (Week 0; Day 0), exam under anesthesia for stem cell coated fistula plug placement Visit 3 (Week 0; Day 1) Visit 4 (Week 2; Month 1) Visit 5 (Week 4; Month 1) Visit 6 (Week 8; Month 2) Visit 7 (Week 12; Month 3) Visit 8 (Week 24; Month 6) Visit 9 (Week 52; Month 12). Visit 10 (Week 104, Month 24)

DETAILED DESCRIPTION:
The Investigators propose to study the safety of autologous mesenchymal stromal cell transfer using a biomatrix (the Gore Bio-A174; Fistula Plug) in a Phase I study using a single dose of 20 million cells. Fifteen adult patients with refractory, rectovaginal fistulizing Crohn's disease will be enrolled. Participants will undergo standard adjuvant therapy including drainage of infection and placement of a draining seton with continuation of pre-existing anti-Crohn's therapy. If the participant is not currently diverted, then participants will undergo a laparoscopic diversion with a loop ileostomy. Six weeks post placement of the draining seton, the seton will be replaced with the MSC loaded Gore Bio-A fistula plug as per current clinical practice. The participants will be subsequently followed for fistula response and closure for 24 months. This is an autologous product derived from the patient and used only for the same patient.

Participants will be screened at outpatient clinic visits and interested qualified participants will be offered participation in the trial and consented. At the first study visit (Visit 1; Screening visit), the patient will be evaluated and assessed. Six weeks post placement of the draining seton, the seton will be replaced with the MSC loaded Gore Bio-A fistula plug. Participants will return on: Day 1, Week 2, Week 4, Week 8, Week 12, Week 24, Week 52, and Week 104.

ELIGIBILITY:
Inclusion Criteria

1. Females 18-65 years of age.
2. Residents of the United States.
3. Crohn's disease with single or multiple draining complex rectovaginal fistulae for at least three months despite standard therapy
4. Concurrent therapies with corticosteroids, 5-ASA drugs, thiopurines, MTX, antibiotics, and anti-TNF therapy are permitted.
5. All patients should have undergone a colonoscopy in last 12 months to rule out malignant or premalignant condition
6. Have no contraindications to MR evaluations: e.g. pacemaker or magnetically active metal fragments, claustrophobia
7. Ability to comply with protocol
8. Competent and able to provide written informed consent
9. Must have failed standard medical therapy including anti-TNF agents
10. Currently with diverting ileostomy or accepting of diverting ileostomy at time of stem cell loaded plug placement.

Exclusion Criteria

1. Inability to give informed consent.
2. Clinically significant medical conditions within the six months before administration of MSCs: e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the patient.
3. Specific exclusions; Evidence of hepatitis B, C, or HIV
4. History of cancer including melanoma (with the exception of localized skin cancers)
5. Investigational drug within thirty (30) days of baseline
6. A resident outside the United States
7. Pregnant or breast feeding.
8. History of clinically significant auto-immunity (other than Crohn's disease) or any previous example of fat-directed autoimmunity
9. Previous allergic reaction to a perianal fistula plug.
10. Allergic to local anesthetics
11. Pregnant patients or trying to become pregnant.
12. entero-vesicular or multiple concurrent perianal tracts

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Rectovaginal fistula, females only eligible
Enrollment: 5 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events (safety and toxicity). | 0-24 months
  Primary Outcome Measure:
  1.Number of participants with treatment-related adverse events (safety and toxicity).
  Participants will have a health assessment and blood work measured at each study visit to monitor for adverse events, such as worsening of the perinal fistulizing disease, abnormal laboratory values, or significant abnormalities in physical examination. The Outcome Measure will be the number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment

SECONDARY OUTCOMES:
Number of participants with response to the treatment regarding potential cessation of drainage from their fistula. | 3-24 months
  Participants will have a clinical assessment of fistula drainage. Participants will be assessed during an office examination if their fistula is draining or not. The Outcome Measure will be the presence or absence of fistula drainage.

CONTACTS AND LOCATIONS:
Overall Officials: Amy L Lightner, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States